CLINICAL TRIAL: NCT02570360
Title: Comparative Effects of Exercise and Treatment-as-usual on Abstinence, Craving, and the Endocannabinoid System in Substance Users
Brief Title: Exercise and Treatment-as-usual in Substance Use Treatment Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0710; 1R36DA040140-01 (NIH); A176000 (Other: UW Madison); EDUC\KINESIOLOGY\KINESIO (Other: UW Madison)
Record Dates: First submitted 2015-09-29; First posted 2015-10-07 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise (Active Comparator): Participants will engage in their outpatient treatment program as-usual, but additionally complete 30mins of moderately intense aerobic exercise 3 times per week for 6 weeks. They will complete 6 weeks of treatment, totaling 18 sessions with exercise.
  Interventions: Behavioral: exercise
- treatment-as-usual (Placebo Comparator): Participants will engage in their outpatient treatment program as-usual,but additionally complete 6 weekly, hour-long visits to complete questionnaires. They will complete 6 weeks of treatment (6 sessions total).
  Interventions: Behavioral: treatment-as-usual

INTERVENTIONS:
Behavioral: exercise — The EX participants will engage in supervised, individual treadmill exercise 3xs/wk at the UW Natatorium. Sessions will consist of a 5-minute warm-up followed by 30 minutes of a moderate to moderately-high intensity exercise and then finish with a 5-minute cool down. Questionnaires will be completed before and after exercise on a weekly basis.
  Arms: exercise
Behavioral: treatment-as-usual — The control (standard care) participants will come to the UW-Natatorium on a weekly basis to complete questionnaires.
  Arms: treatment-as-usual

SUMMARY:
The research study compares the substance abuse treatment outcomes (e.g., craving, withdrawal symptoms, rates of use, abstinence) of standard intensive outpatient care, with or without an added 6-wk aerobic exercise component. In addition, certain biomarkers associated with both exercise and substance use (e.g., endocannabinoids and cortisol) will be assessed. In a rolling admissions format over the course of a year, approximately 36 treatment-seeking substance users who are currently receiving Intensive Outpatient Treatment through a local Alcohol or Other Drug Abuse agency will be randomized to either receive 6 weeks aerobic exercise training in addition to standard care or standard care with 6 weekly laboratory visits to complete questionnaires (18 per group).

ELIGIBILITY:
Inclusion Criteria:

* Intact cognitive status and ability to provide informed consent
* ability to read and write in English sufficient to provide consent and complete study questionnaires
* current diagnosis of a single or of multiple substance use disorders
* currently enrolled in an Intensive Outpatient Treatment substance use program
* desire to quit and to seek treatment for substance use
* currently sedentary, not participating in any formal/structured exercise program

Exclusion Criteria:

* a history or present diagnosis of severe depression, psychotic, or bipolar disorder
* presence of cardiac disease or any other medical condition that would make engaging in exercise unsafe
* Undergoing methadone treatment
* chronic conditions such as cancer, diabetes, kidney disease, or autoimmune disorders
* women who are pregnant or planning to become pregnant

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Withdrawal Checklist: Change in physical and psychological withdrawal symptoms over the course of the intervention | up to 6 weeks
  withdrawal symptoms will be assessed using the Withdrawal Checklist which asks participants to rate the severity of a variety physical and psychological symptoms over the past 48 hours. The total score on the Withdrawal Checklist will be used to provide an overall measured of withdrawal.

SECONDARY OUTCOMES:
change in cortisol concentrations | measured before and after sessions (via saliva swab) during the first, third, and sixth weeks of the 6-week intervention
change in endocannabinoid concentrations | measured before and after sessions (via single venipuncture)during the first, third, and sixth weeks of the 6-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Angelique Brellenthin, MS, Principal Investigator — UW-Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

REFERENCES:
- [Result] Brellenthin AG, Crombie KM, Hillard CJ, Brown RT, Koltyn KF. Psychological and endocannabinoid responses to aerobic exercise in substance use disorder patients. Subst Abus. 2021;42(3):272-283. doi: 10.1080/08897077.2019.1680480. Epub 2019 Nov 15. PMID 31729933